CLINICAL TRIAL: NCT00158067
Title: Automated Response to Spontaneous Epileptiform Activity Using the External Responsive Neurostimulator (eRNS) System Clinical Investigation
Brief Title: Study of an External Responsive Neurostimulator System on Epileptiform Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroPace (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1006633
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; Neurostimulation
MeSH Terms: conditions — Epilepsy | interventions — Drug Delivery Systems

INTERVENTIONS:
Device: external Responsive Neurostimulator (eRNS) System

SUMMARY:
This feasibility clinical investigation is designed to demonstrate that the NeuroPace external Responsive Neurostimulator (model eRNS-300) can safely deliver responsive electrical stimulation automatically to affect epileptiform activity. The eRNS-300 is based on an implantable neurostimulator that has been adapted for acute, external use in a hospital setting.

DETAILED DESCRIPTION:
The Automated Response to Spontaneous Epileptiform Activity using the External Responsive Neurostimulator (eRNS) system clinical investigation involves subjects who are undergoing intracranial monitoring for the evaluation of epilepsy surgery and who are being monitored in the hospital's epilepsy monitoring unit. During the subject's participation, at the discretion of the investigator, the subject will be connected to the eRNS. The eRNS is an investigational device that attaches to standard intracranial electrode monitoring equipment to monitor the subject's seizure activity. It is anticipated that the subject may be connected to the eRNS for a period of time extending from one day to a few weeks. After the subject has enough seizures to complete their evaluation for epilepsy surgery, the physician may enable the responsive stimulation settings for the eRNS. The subject's participation in the clinical investigation will be complete prior to the removal of their intracranial electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing evaluation for epilepsy surgery in a manner consistent with the Surgery for Epilepsy, NIH Consensus Statement, 1990 Mar 19-21; 8(2); 1-20.
* Subject is implanted with intracranial electrodes.
* Subject is under constant medical supervision while implanted with the intracranial electrodes.
* Subject is twelve (12) years of age or older.

Exclusion Criteria:

* Subject is pregnant.
* Subject has a clinically significant or unstable medical condition that, in the opinion of the investigator, would make it inadvisable for the individual to participate.
* Subject has a progressive central nervous system disease or serious acute or ongoing systemic illnesses.
* Subject has an active psychosis, severe depression, suicidal ideation or psychiatric conditions associated with impaired judgment.
* Subject is considered at high risk, for any reason, by any of the investigators.
* Subject is implanted with a medical device that might interfere with the eRNS. (This includes, but is not limited to direct brain neurostimulators, pacemakers, implantable cardiac defibrillators, spinal cord stimulators, vagal nerve stimulators, cochlear implants)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-03; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Scottsdale, Arizona
  - Research Site, Augusta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York